CLINICAL TRIAL: NCT00595777
Title: Does the Institutionalisation of Pain Assessment Using the EPAT© Package Reduce the Pain in Cancer In-patients More Than Usual Care; a Cluster Randomised Trial.
Brief Title: Edinburgh Pain Assessment Tool (EPAT©) Study
Acronym: EPAT©
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 06/MRE10/84
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Cancer
Keywords: Institutional change; Improved pain management
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Comparison (No Intervention): The centres allocated to the comparison group will continue to provide usual care only.
- 2. Experimental (Experimental): The EPAT package consists of an educational programme, which deals with the common barriers to effective cancer pain control and the bedside pain tool.
  Interventions: Behavioral: EPAT© Educational Package

INTERVENTIONS:
Behavioral: EPAT© Educational Package — The EPAT package consists of an education programme, which deals with the known common barriers to effective pain control and the bedside pain tool. The pain tool is uniquely incorporated into the vital signs chart to enable a systematic approach to cancer pain assessment and review. EPAT consists of 2 steps: step 1 is a colour-coded pain assessment on the bedside vital signs chart. Patients with moderate or severe pain on step 1 will progress to to step 2, which helps to identify the aetiology of the pain, screening for opioid side effects and is linked via flags to simple management plans. The intervention will be delivered to the clusters randomised to the intervention, after collection of baseline data (pre-intervention data) on 50 patients.
  Arms: 2. Experimental

SUMMARY:
To determine if the institutionalisation of a regular systematic approach to the assessment of pain in inpatient cancer units using the Edinburgh Pain Assessment Tool (EPAT©) leads to better control of pain than that achieved by usual care.

DETAILED DESCRIPTION:
Background and relevance to cancer - Pain associated with cancer has a severe negative impact on quality of life and can also limit a patient's ability to tolerate potentially life-saving tumoricidal treatment. Unfortunately in practice only half of cancer patients receive adequate pain control. A fundamental reason for this is inadequate assessment of pain. The institutionalisation of pain assessment as a 5th vital sign on the bedside chart combined with training and guidance in pain management (EPAT) is a potentially effective solution.

We have already evaluated the feasibility and efficacy of EPAT in a randomised trial of 150 oncology inpatients and found that by Day 4 after admission 90% reported adequate pain control compared to only 52% of those who received usual care.

Aims - We now want to evaluate the effectiveness and cost-effectiveness of EPAT in practice and ask: Does it reduce cancer pain more that usual care? Are there adverse effects? Is it cost effective?

Outline plan - A UK-wide cluster randomised controlled trial of 18 inpatient cancer centres of which half will use the EPAT package and half usual care. The trial outcomes are clinically significant improvement, adverse effects such as opiate toxicity and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Able and consent to complete a Brief Pain Inventory score
* Aged over 18 years
* Have a pain score equal to or greater than 4 out of 10 at first assessment point (within 24 hours of admission) and pain is cancer related
* Are expected to be available for pain assessment at 3 days after admission

Exclusion Criteria:

* Do not consent to take part in the study or who are too ill to take part, including those with severe mental health problems
* Do not have cancer-related pain
* Are under 18 years of age
* Have a pain score of less than 4
* Are not expected to be available for pain assessment at 3 days after admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1928 (Actual)
Dates: Start 2007-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The magnitude of change in pain scores at the 2 evaluation points measured by patient self-rating | Maximum study duration is 9 days per patient

SECONDARY OUTCOMES:
Magnitude of change in BPI scores over the 2 evaluation points (includes impact on function) | Maximum study duration is 9 days per patient
Patient satisfaction with attention to pain | Maximum study duration is 9 days per patient
Global distress | Maximum study duration is 9 days per patient

CONTACTS AND LOCATIONS:
Overall Officials: Marie Fallon, Study Director — University of Edinburgh; Michael Sharpe, Study Director — University of Edinburgh; Lesley Colvin, Study Director — University of Edinburgh; Gordon Murray, Study Director — University of Edinburgh
Locations (19):
- United Kingdom (19):
  - Mount Vernon Cancer Centre, Northwood, Middlesex
  - Bristol Haematology and Oncology Centre, Bristol, Sommerset
  - Belfast City Hospital, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Addenbrookes Hospital, Cambridge
  - Velindre Hospital, Cardiff
  - The Western General Hospital, Edinburgh
  - Beaston Oncology Centre, Glasgow
  - Hull Royal Infirmary, Hull
  - St. James's Hospital, Leeds
  - Clatterbridge Centre for Oncology, Liverpool
  - The Royal Marsden Hospital, London
  - The Christie, Manchester
  - Freeman Hospital, Newcastle
  - City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Southampton University Hospital, Southampton
  - The Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] Fallon M, Walker J, Colvin L, Rodriguez A, Murray G, Sharpe M; Edinburgh Pain Assessment and Management Tool Study Group. Pain Management in Cancer Center Inpatients: A Cluster Randomized Trial to Evaluate a Systematic Integrated Approach-The Edinburgh Pain Assessment and Management Tool. J Clin Oncol. 2018 May 1;36(13):1284-1290. doi: 10.1200/JCO.2017.76.1825. Epub 2018 Mar 15. PMID 29543567